CLINICAL TRIAL: NCT01176240
Title: A Multi-center, Double-blind, Randomized, Parallel-Group, Placebo-Controlled Study to Assess the Clinical Effect of Droxidopa in the Treatment of Symptomatic Neurogenic Orthostatic Hypotension in Patients With Parkinson's Disease
Brief Title: A Two Part Study (306A/306B) to Assess Droxidopa in Treatment of NOH in Patients With Parkinson's Disease
Acronym: 306A/306B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chelsea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Droxidopa NOH306 (306A / 306B)
Record Dates: First submitted 2010-07-30; First posted 2010-08-05 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-04

CONDITIONS: Orthostatic Hypotension; Parkinson's Disease
Keywords: lightheadedness; unsteadiness; dizziness; weak; fatigue; concentration; head & neck pain; standing/walking for a short time; standing/walking for a long time; Neurogenic Orthostatic Hypotension; falls; NOH; Parkinson's disease; weakness
MeSH Terms: conditions — Hypotension, Orthostatic; Parkinson Disease; Dizziness; Asthenia; Fatigue; Neck Pain | interventions — Droxidopa; Mannitol; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Droxidopa (Experimental): droxidopa active drug
  Interventions: Drug: Droxidopa
- Placebo (Placebo Comparator): Placebo matched control
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Droxidopa — 100 mg and 200 mg capsules 100, 200, 300, 400, 500, 600mg TID dosing for up to 8 weeks of treatment
  Other Names: Northera; L-DOPS; L-threo-dihydroxyphenylserine; SM-5688
  Arms: Droxidopa
Other: Placebo — Placebo
  Other Names: Mannitol, Sugar Pill
  Arms: Placebo

SUMMARY:
This is a study to evaluate the effects of an investigational drug, Droxidopa, in participants with neurogenic orthostatic hypotension (NOH), associated with Parkinson's disease. Droxidopa is being studied to determine the effects on blood pressure changes upon standing up (orthostatic challenge). Symptoms and activity measurements, including patient reported falls, will be evaluated to determine the effectiveness of the study drug.

Symptoms of NOH may include any of the following:

* Dizziness, light-headedness, feeling faint or feeling like you may blackout
* Problems with vision (blurring, seeing spots, tunnel vision, etc.)
* Weakness
* Fatigue
* Trouble concentrating
* Head & neck discomfort (the coat hanger syndrome)
* Difficulty standing for a short time or a long time
* Trouble walking for a short time or a long time

The study duration is a maximum of approximately 14 weeks including up to 2 weeks for screening, up to 2 weeks for proper dose finding, followed by an 8 week treatment period and a follow-up visit after 2 weeks. A sufficient number of patients will be screened to allow approximately 211 randomized patients. An extension study is also available to continue treatment if determined appropriate by the study doctor. This Study is NCT01132326 sponsored by Chelsea Therapeutics and is enrolling by invitation only.

DETAILED DESCRIPTION:
Systolic blood pressure is transiently and minimally decreased in healthy individuals upon standing. Normal physiologic feedback mechanisms work through neurally-mediated pathways to maintain the standing blood pressure, and thus maintain adequate cerebral perfusion. The compensatory mechanisms that regulate blood pressure upon standing are dysfunctional in subjects with orthostatic hypotension (OH), a condition that may lead to inadequate cerebral perfusion with accompanying symptoms of syncope, dizziness or lightheadedness, unsteadiness and blurred or impaired vision, among other symptoms.

Orthostatic hypotension may be a severely disabling condition which can seriously interfere with the quality of life of afflicted subjects. Currently available therapeutic options provide some symptomatic relief in a subset of subjects, but are relatively ineffective and are often accompanied by severe side effects that limit their usefulness. Support garments (tight-fitting leotard) may prove useful in some subjects, but is difficult to don without family or nursing assistance, especially for older subjects. Midodrine, fludrocortisone, methylphenidate, ephedrine, indomethacin and dihydroergotamine are among some of the pharmacological interventions that have been used to treat orthostatic hypotension, although only midodrine is specifically approved for this indication. The limitations of these currently available therapeutic options, and the incapacitating nature and often progressive downhill course of disease, point to the need for an improved therapeutic alternative.

Symptomatic OH in patients with Parkinson's disease is thought to be a consequence of norepinephrine depletion leading to low systolic blood pressure (SBP) and cerebral-hypoperfusion (reduced blood flow to the brain). Therapy with droxidopa results in increased levels of norepinephrine which should lead to improved SBP and cerebral perfusion thereby reducing the signs and symptoms of NOH. The present study will evaluate the clinical benefit in NOH patients with PD treated with droxidopa compared to those treated with placebo.

Participation in the study will last a maximum of 14 weeks consisting of a 2 week (maximum) screening/baseline period; a 2 week (maximum) double-blind dose titration; an 8 week double-blind placebo-controlled treatment period; and a 2 week follow-up period. An extension study is also available to continue treatment if determined appropriate by the study doctor. This Study is NCT01132326 sponsored by Chelsea Therapeutics and is enrolling by invitation only.

Droxidopa:

Droxidopa [also, known as L-threo-3,4-dihydroxyphenylserine, L-threo-DOPS, or L-DOPS] is the International non-proprietary name (INN) for a synthetic amino acid precursor of norepinephrine (NE), which was originally developed by Sumitomo Pharmaceuticals Co., Limited, Japan. It has been approved for use in Japan since 1989. Droxidopa has been shown to improve symptoms of orthostatic hypotension that result from a variety of conditions including Shy Drager syndrome (Multiple System Atrophy), Pure Autonomic Failure, and Parkinson's disease. There are four stereoisomers of DOPS; however, only the L-threo-enantiomer (droxidopa) is biologically active. Stereoisomers and enantiomers are compounds that have the same chemical elements; however, they may react differently as the elements are positioned in different locations.

The exact mechanism of action of droxidopa in the treatment of symptomatic NOH has not been precisely defined; however, its NE replenishing properties with concomitant recovery of decreased noradrenergic activity are considered to be of major importance.

Droxidopa has been marketed in Japan since 1989. Data from clinical studies and post-marketing surveillance programs conducted in Japan show that the most commonly reported adverse drug reactions with droxidopa are increased blood pressure, nausea, and headache. In clinical studies, the prevalence and severity of droxidopa adverse effects appear to be similar to those reported by the placebo control arm.

ELIGIBILITY:
Inclusion criteria:

1. 18 years or over
2. Clinical diagnosis of Parkinson's disease
3. Clinical diagnosis of symptomatic neurogenic orthostatic hypotension

At their baseline visit (Visit 2), patients must demonstrate:

* a score of at least 3 or greater on the OHQ composite
* a score of at least 3 or greater on the clinician CGI-S
* a fall of at least 20 mmHg in their systolic blood pressure, or 10 mmHg in their diastolic blood pressure, within 3 minutes of standing 4. Provide written informed consent to participate in the study and understand that they may withdraw their consent at any time without prejudice to their future medical care

Exclusion Criteria:

1. Score of 23 or lower on the mini-mental state examination (MMSE)
2. Concomitant use of vasoconstricting agents for the purpose of increasing blood pressure;

   - Patients taking vasoconstricting agents such as ephedrine, dihydroergotamine, or midodrine must stop taking these drugs at least 2 days or 5 half-lives (whichever is longer) prior to their baseline visit (Visit 2) and throughout the duration of the study
3. Concomitant use of anti-hypertensive medication for the treatment of essential hypertension
4. Have changed dose, frequency or type of prescribed medication, within two weeks of baseline visit (Visit 2) with the following exceptions:

   * Vasoconstricting agents such a ephedrine, dihydroergotamine, or midodrine
   * Short courses (less than 2 weeks) of medications or treatments that do not interfere with, or exacerbate the patient's condition under study (e.g. antibiotics)
5. Known or suspected alcohol or substance abuse within the past 12 months (DSM-IV definition of alcohol or substance abuse)
6. Women who are pregnant or breastfeeding
7. Women of child bearing potential (WOCP) who are not using at least one method of contraception with their partner
8. Male patients who are sexually active with a woman of child bearing potential (WOCP) and not using at least one method of contraception
9. Untreated closed angle glaucoma, or treated closed angle glaucoma that, in the opinion of an ophthalmologist, might result in an increased risk to the patient
10. Sustained severe hypertension (BP ≥ 180 mmHg systolic or ≥ 110 mmHg diastolic in the seated or supine position which is observed in 3 consecutive measurements over an hour)
11. Any significant uncontrolled cardiac arrhythmia
12. History of myocardial infarction, within the past 2 years
13. Current unstable angina
14. Congestive heart failure (NYHA Class 3 or 4)
15. Diabetic autonomic neuropathy
16. History of cancer within the past 2 years other than a successfully treated, non-metastatic cutaneous squamous cell or basal cell carcinoma or cervical cancer in situ
17. Gastrointestinal condition, which in the Investigator's judgment, may affect the absorption of study drug (e.g. ulcerative colitis, gastric bypass)
18. Any major surgical procedure within 30 days of the baseline visit (Visit 2)
19. Previously treated with droxidopa
20. Currently receiving any investigational drug or have received an investigational drug within 30 days of the baseline visit (Visit 2)
21. Any condition or laboratory test result, which in the Investigator's judgment, might result in an increased risk to the patient, or would affect their participation in the study. Additionally the Investigator has the ability to exclude a patient if for any reason they feel the subject is not a good candidate for the study or will not be able to follow study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2010-06; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hauser, M.D., Principal Investigator — University of South Florida; Lawrence A. Hewitt, Ph.D., Study Chair — Chelsea Therapeutics, Inc.; William Schwieterman, M.D., Study Director — Chelsea Therapeutics, Inc.
Locations (60):
- United States (60):
  - Neurology Neurodiagnostic Lab, Alabaster, Alabama
  - Neurological Physicians of Arizona, Gilbert, Arizona
  - Xenoscience, Phoenix, Arizona
  - Barrow Neurology Clinic, Phoenix, Arizona
  - Banner Health, Sun City, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Northwest Neuro Specialists P.L.L.C., Tucson, Arizona
  - Caring Clinical Research Incorporated, Laguna Hills, California
  - Hoag Memorial Hospital, Presbyterian, Newport Beach, California
  - Neurosearch - Pasadena, Pasadena, California
  - Alliance Clinical Research, LLC, Poway, California
  - Neurosearch, Inc., Reseda, California
  - Neurosearch II, Inc., Ventura, California
  - Neurology Consultants Medical Group, Whittier, California
  - Associated Neurologist of Southern Connecticut, PC, Fairfield, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Eastern Connecticut Neurology Specialists, Manchester, Connecticut
  - Parkinson's Disease & Movement Disorder Disoder, Boca Raton, Florida
  - Pharmax Research Clinic, LLC, Miami, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Neurostudies Inc., Port Charlotte, Florida
  - Parkinson's Disease Treatment Center of Southwest Florida, Port Charlotte, Florida
  - Lovelace Scientific Research, Sarasota, Florida
  - Tampa General University of South Florida, Tampa, Florida
  - Vero Neurology, Vero Beach, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Neurology Specialists of Decatur Research Center, Decatur, Georgia
  - Prism Research Group, Rome, Georgia
  - Alexian Brothers Hospital Network, Elk Grove Village, Illinois
  - Precise Clinical Research, Topeka, Kansas
  - North Oaks Health System, Hammond, Louisiana
  - Harvard Vanguard Medical Associates, Boston, Massachusetts
  - Detroit Clinical Research Center, Novi, Michigan
  - Northern Michigan Neurology, Traverse City, Michigan
  - Gulf Coast Neurology Center, PLLC, Ocean Springs, Mississippi
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Wellness and Research Center, Belvidere, New Jersey
  - AdvanceMed Research, Lawrenceville, New Jersey
  - Shore Neurology, Toms River, New Jersey
  - Upstate Clinical Research, LLC, Albany, New York
  - David L. Kreitzman, M.D., PC, Commack, New York
  - Kingston Neurological Associates, Kingston, New York
  - Parker Jewish Institute For Health Care and Rehabilitation Foundation, New Hyde Park, New York
  - Beth Israel Medical Center, New York, New York
  - New York University, New York, New York
  - Neurological Care of CNY, Syracuse, New York
  - Asheville Neurology Specialists, PA, Asheville, North Carolina
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - Clinical Trials of America Inc, Winston-Salem, North Carolina
  - Community Research, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Toledo, Toledo, Ohio
  - Movement Disorder Clinic of Oklahoma PLLC, Tulsa, Oklahoma
  - Ilumina Clinical Associates, Johnstown, Pennsylvania
  - Clinical Trials Research Services LLC, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - JM Neuroscience Research, Salt Lake City, Utah
  - Neurological Associates, Inc., Richmond, Virginia
  - Sentara Neurology Specialists, Virginia Beach, Virginia

REFERENCES:
- [Background] Birkmayer W, Birkmayer G, Lechner H, Riederer P. DL-3,4-threo-DOPS in Parkinson's disease: effects on orthostatic hypotension and dizziness. J Neural Transm. 1983;58(3-4):305-13. doi: 10.1007/BF01252816. PMID 6420517
- [Background] Movement Disorder Society Task Force on Rating Scales for Parkinson's Disease. The Unified Parkinson's Disease Rating Scale (UPDRS): status and recommendations. Mov Disord. 2003 Jul;18(7):738-50. doi: 10.1002/mds.10473. PMID 12815652
- [Background] Goldstein DS, Pechnik S, Holmes C, Eldadah B, Sharabi Y. Association between supine hypertension and orthostatic hypotension in autonomic failure. Hypertension. 2003 Aug;42(2):136-42. doi: 10.1161/01.HYP.0000081216.11623.C3. Epub 2003 Jun 30. PMID 12835329
- [Background] Kachi T, Iwase S, Mano T, Saito M, Kunimoto M, Sobue I. Effect of L-threo-3,4-dihydroxyphenylserine on muscle sympathetic nerve activities in Shy-Drager syndrome. Neurology. 1988 Jul;38(7):1091-4. doi: 10.1212/wnl.38.7.1091. PMID 3133573
- [Background] Kaufmann H, Saadia D, Voustianiouk A, Goldstein DS, Holmes C, Yahr MD, Nardin R, Freeman R. Norepinephrine precursor therapy in neurogenic orthostatic hypotension. Circulation. 2003 Aug 12;108(6):724-8. doi: 10.1161/01.CIR.0000083721.49847.D7. Epub 2003 Jul 28. PMID 12885750
- [Background] Yanagisawa N, Ikeda S, Hashimoto T, Hanyu N, Nakagawa S, Fujimori N, Ushiyama M. [Effects of L-threo-Dops on orthostatic hypotension in Parkinson's disease]. No To Shinkei. 1998 Feb;50(2):157-63. Japanese. PMID 9513205
- [Background] Malamut, R., Freeman, R., Gilden, J., Tulloch, J., Kaufmann, H., 2005. A multi-center, double-blind, randomized, placebo controlled, cross-over study to assess the clinical benefit of midodrine in patients with neurogenic orthostatic hypotension. Clin. Auto. Res. 15 (5) 337[abstract].
- [Background] Narabayashi, H., Nakanishi, T., Kanazawa, I., Yoshida, M., Mizuno, Y., Yanagisawa, N., Kondo, T. 1987. Clinical effects of L-threo-3,4-dihydroxyphenylserine in Parkinson's disease and Parkinson syndrome: Results of multi-center open study at 45 institutions. Yakuri To Chiryo (Jpn. Pharmacol. Ther.) 15(Suppl. 2):411 to 443.
- [Background] Sobue, I., Senda, Y., Suzuki, T., Narabayashi, I., Hirayama, K. 1987. Clinical effects of L-threo-3,4-dihydroxyphenylserine on orthostatic hypotension in Shy-Drager Syndrome and its related diseases. Shinkei Naika Chiryo [Neurol. Ther.] 4(2):199-208.
- [Derived] Heller GZ, Couturier DL, Heritier SR. Beyond mean modelling: Bias due to misspecification of dispersion in Poisson-inverse Gaussian regression. Biom J. 2019 Mar;61(2):333-342. doi: 10.1002/bimj.201700218. Epub 2018 Jul 12. PMID 30003579
- [Derived] Biaggioni I, Arthur Hewitt L, Rowse GJ, Kaufmann H. Integrated analysis of droxidopa trials for neurogenic orthostatic hypotension. BMC Neurol. 2017 May 12;17(1):90. doi: 10.1186/s12883-017-0867-5. PMID 28494751
- [Derived] Francois C, Rowse GJ, Hewitt LA, Vo P, Hauser RA. Analysis of number needed to treat for droxidopa in patients with symptomatic neurogenic orthostatic hypotension. BMC Neurol. 2016 Aug 18;16(1):143. doi: 10.1186/s12883-016-0665-5. PMID 27538531
- [Derived] Hauser RA, Hewitt LA, Isaacson S. Droxidopa in patients with neurogenic orthostatic hypotension associated with Parkinson's disease (NOH306A). J Parkinsons Dis. 2014;4(1):57-65. doi: 10.3233/JPD-130259. PMID 24326693

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Post-randomization, up to 2 weeks dose titration followed by 8 wks at optimal dose.
  The first 51 patients enrolled in the study were analyzed as a separate group in an interim analysis (Study 306A).
  The final 171 patients remained blinded until the end of the study and analyzed as a separate study (Study 306B).
Period: Study 306A
Arm/Group | Droxidopa | Placebo
Started | 24 | 27
Completed | 21 | 24
Not Completed | 3 | 3
Not completed — Lack of Efficacy | 2 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Stop due to diverse problems | 1 | 0
Period: Study 306B
Arm/Group | Droxidopa | Placebo
Started | 89 | 85
Took at Least 1 Dose of Study Drug | 87 (Two randomized patients discontinued before receiving study drug.) | 84 (One randomized patient discontinued before receiving study drug.)
1 wk of Stable Dosing and Visit 4 | 69 | 78
2 wk of Stable Dosing and Visit 5 | 68 | 75
4 wk of Stable Dosing and Visit 6 | 67 | 73
Completed | 63 | 68
Not Completed | 26 | 17
Not completed — Lack of Efficacy | 5 | 3
Not completed — Adverse Event | 10 | 5
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Supine Hypertension | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — withdrew prior to dosing | 2 | 1

BASELINE CHARACTERISTICS:
Population: The population only includes those patients who were randomized and took at least one dose of study drug (n=222).
  The first 51 patients enrolled in the study were analyzed as a separate group in an interim analysis (Study 306A).
  The final 171 patients remained blinded until the end of the study and analyzed as a separate study (Study 306B).
Groups:
- Study 306A: Droxidopa; Study 306B: Droxidopa: droxidopa active drug
  Droxidopa: 100 mg and 200 mg capsules 100, 200, 300, 400, 500, 600mg TID dosing for up to 8 weeks of treatment
- Study 306A: Placebo; Study 306B: Placebo: Placebo matched control
  Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Study 306A: Droxidopa | Study 306A: Placebo | Study 306B: Droxidopa | Study 306B: Placebo | Total
Number analyzed (Participants) | 24 | 27 | 87 | 84 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (7.30) | 72.9 (7.76) | 72.5 (7.64) | 72.2 (7.97) | 72.4 (7.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 27 | 30 | 77
  Male | 14 | 17 | 60 | 54 | 145
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 1 | 5
  White | 24 | 25 | 84 | 83 | 216
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 27 | 87 | 84 | 222

OUTCOME MEASURES:

1. Primary Outcome: 306A Efficacy: Change in Orthostatic Hypotension Questionnaire Score (OHQ)
Description: The primary efficacy endpoint for 306A is the relative mean change in Orthostatic Hypotension Questionnaire (OHQ) composite score from baseline to end of study. The OHQ is the average of two sub-scales, the Orthostatic Hypotension Symptom Assessment Scale (OHSA) and the Orthostatic Hypotension Daily Activities Scale (OHDAS). Each asks the patient to rate their symptoms or disease impact over the past week. The OHSA sub-scale is the average of six items: 1) Dizziness, lightheadedness, feeling faint or feeling like you might black out; 2) Problems with vision; 3) Weakness; 4) Fatigue; 5) Trouble concentrating; and 6) Head/neck discomfort. The OHDAS sub-scale is the average of four items: 1) Standing for a short time; 2) Standing for a long time; 3) Walking for a short time; and 4) Walking for a long time. Each item is scored on a Likert scale from 0 to 10, with 10 being the most severe.
  For the change from baseline, negative numbers represent improvement from baseline in OHQ score.
Time Frame: Baseline, Week 8
Population: LOCF was used to impute values for patients who did not have an end of study visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 24 | 27
units on a scale | -2.2 (2.44) | -2.1 (2.49)
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Study 306A was initially designed as a blinded interim analysis by an independent DMC to ensure that the overall study was adequately powered. Study 306A was not powered to provide statistical significance as a stand alone study. Thus, no additional efficacy end points were prospectively defined beyond the primary end point; Test type: Superiority or Other; p = 0.978, ANCOVA; ANCOVA model that includes treatment as a factor and baseline OHQ composite score as a co-variate

2. Primary Outcome: 306B Efficacy: Change in Dizziness/Lightheadedness/Feeling Faint/Feeling Like You Might Black Out (OHSA Item 1)
Description: OHSA item 1 scale range: 0 (none) -10 (worst), likert scale. Change: score at Week 1 minus score at baseline. A negative score indicates an improvement in symptoms during the double-blind randomized phase relative to value at baseline.
Time Frame: Baseline, Week1
Population: The primary analysis was defined as those patients who completed 1 week of dosing at the identified optimal dose of study medication and completed the visit 4 (1 week) efficacy evaluation. Patients who did not have week 1 efficacy data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 69 | 78
units on a scale | -2.3 (2.95) | -1.3 (3.16)
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.018, Mantel Haenszel — Statistical analysis plan involved a hierarchical assessment of secondary endpoints to prevent inflation of type I errors; Mantel-Haenszel statistic comparing treatment groups based on rank statistics adjusted for the covariate OHSA Item 1 value at baseline

3. Post Hoc Outcome: 306A Efficacy: Patient Reported Falls
Description: The total number of patient reported falls during the 8 week treatment period
Time Frame: Baseline, Week 8
Measure: Number; unit: total falls per group
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 24 | 27
total falls per group | 79 | 192

4. Secondary Outcome: 306B Efficacy: Change in OHSA Item 1 From Baseline to Week 2 (Visit 5)
Description: OHSA item 1 scale range: 0 (none) -10 (worst), likert scale. Change: score at Week 2 minus score at baseline. A negative score indicates an improvement in symptoms during the double-blind randomized phase relative to value at baseline.
Time Frame: Baseline, Week2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 68 | 75
units on a scale | -1.9 (2.86) | -1.6 (2.97)
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.60, Wilcoxon (Mann-Whitney) — Statistical analysis plan involved a hierarchical assessment of secondary endpoints to prevent inflation of type I errors. As the first secondary endpoint was not positive, statistical analysis was not performed on additional secondary endpoints; [statistical method as in outcome 2, analysis 1]

5. Secondary Outcome: 306B Efficacy: Change in OHSA Item 1 From Baseline to Week 4 (Visit 6)
Description: OHSA item 1 scale range: 0 (none) -10 (worst), likert scale. Change: score at Week 4 minus score at baseline. A negative score indicates an improvement in symptoms during the double-blind randomized phase relative to value at baseline.
Time Frame: Baseline, Week4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 67 | 73
units on a scale | -2.0 (3.08) | -1.5 (2.74)

6. Secondary Outcome: 306B Efficacy: Change in Systolic Blood Pressure (SBP) Measurements Post Standing From Baseline to Week 1
Description: Measure: Lowest standing systolic blood pressure reading of immediately post standing and 3 minutes post standing. Change: standing systolic blood pressure at Week 1 (Visit 4) minus standing systolic blood pressure at baseline. A positive score indicates an improvement in standing systolic blood pressure during the double-blind randomized phase relative to value at baseline.
Time Frame: Baseline, Week 1
Population: One droxidopa patient did not complete the standing blood pressure measurements of the orthostatic standing test at visit 4 (one week of stable dosing)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 68 | 78
mmHg | 6.4 (18.85) | 0.7 (20.18)

7. Secondary Outcome: 306B Efficacy: Change in OHSA Item 1 From Baseline to Week 8 (Visit 7)
Description: OHSA item 1 scale range: 0 (none) -10 (worst), likert scale. Change: score at Week 8 minus score at baseline. A negative score indicates an improvement in symptoms during the double-blind randomized phase relative to value at baseline.
Time Frame: Baseline, Week 8
Population: The analysis was defined as those patients who completed 8 week of dosing and completed the visit 7 (8 week) efficacy evaluation. Patients who did not have week 8 efficacy data were excluded from the analysis. Of note, 2 patients completed the 8 week double blind study, but did not complete the efficacy evaluations at the final visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 63 | 68
units on a scale | -2.1 (3.03) | -1.5 (2.91)

8. Secondary Outcome: 306B Efficacy: Rate of Patient Reported Falls
Description: The average number of patient reported falls per week.
Time Frame: up to 10 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: falls per week
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 69 | 78
falls per week | 0.4 (0.84) | 2.0 (12.95)

9. Secondary Outcome: 306B Efficacy: Change in Orthostatic Hypotension Questionnaire Score (OHQ)
Description: The relative mean change in Orthostatic Hypotension Questionnaire (OHQ) composite score from baseline to end of study. The OHQ is the average of two sub-scales, the Orthostatic Hypotension Symptom Assessment Scale (OHSA) and the Orthostatic Hypotension Daily Activities Scale (OHDAS). Each asks the patient to rate their symptoms or disease impact over the past week. The OHSA sub-scale is the average of six items: 1) Dizziness, lightheadedness, feeling faint or feeling like you might black out; 2) Problems with vision; 3) Weakness; 4) Fatigue; 5) Trouble concentrating; and 6) Head/neck discomfort. The OHDAS sub-scale is the average of four items: 1) Standing for a short time; 2) Standing for a long time; 3) Walking for a short time; and 4) Walking for a long time. Each item is scored on a Likert scale from 0 to 10, with 10 being the most severe.
  For the change from baseline, negative numbers represent improvement from baseline in OHQ score.
Time Frame: Baseline, Week 8
Population: The primary analysis was defined as those patients who completed 8 week of dosing and completed the visit 7 (8 week) efficacy evaluation. Patients who did not have week 8 efficacy data were excluded from the analysis. Of note, 2 patients completed the 8 week double blind study, but did not complete the efficacy evaluations at the final visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 63 | 68
units on a scale | -2.2 (2.29) | -2.0 (2.18)

10. Post Hoc Outcome: Study 306A: Change in Dizziness/Lightheadedness/Feeling Faint/Feeling Like You Might Black Out (OHSA Item 1) From Baseline to Week 1
Description: OHSA item 1 scale range: 0 (none) -10 (worst), likert scale. Change: score at Week 1 minus score at baseline. A negative score indicates improvement in symptoms during the double-blind randomized phase relative to value at baseline.
Time Frame: Baseline, Week 1
Population: Last observation carried forward was used to impute missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 24 | 27
units on a scale | -3.1 (3.39) | -1.6 (3.12)
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.238, ANCOVA; ANCOVA model that includes treatment as a factor and baseline OHQ composite score as a co-variate

ADVERSE EVENTS:
Description: Subjects with more than 1 of a given AE, the subject is counted only once for that AE. Subject with more than one AE in a system organ class (SOC), the subject is counted only once in that SOC.
  Only dosed patients included in Safety Set.
  Droxidopa Safety Set includes 3 patients randomized to placebo who were mistakenly dosed with droxidopa.
Groups:
- Droxidopa: droxidopa active drug
  Droxidopa: 100 mg and 200 mg capsules 100, 200, 300, 400, 500, 600mg TID dosing for up to 8 weeks of treatment
  Droxidopa Safety set includes 3 patients randomized to placebo who were mistakenly dosed with droxidopa for short periods of time during the trial.
- Placebo: Placebo matched control
  Placebo: Placebo
  Placebo Safety set excludes 3 patients randomized to placebo who were mistakenly dosed with droxidopa for short periods of time during the trial.
Arm/Group | Droxidopa | Placebo
Serious Adverse Events (participants affected / at risk) | 5/114 | 4/108
Other Adverse Events (participants affected / at risk) | 54/114 | 52/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Droxidopa (N=114) | Placebo (N=108)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Droxidopa (N=114) | Placebo (N=108)
Headache (Nervous system disorders) | 15 (19) | 8 (8)
Dizziness (Nervous system disorders) | 11 (13) | 5 (6)
Nausea (Gastrointestinal disorders) | 10 (13) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 8 (9)
Fatigue (General disorders) | 8 (8) | 6 (7)
Oedema peripheral (General disorders) | 5 (5) | 6 (6)
Contusion (Injury, poisoning and procedural complications) | 6 (7) | 12 (14)
Excoriation (Injury, poisoning and procedural complications) | 6 (6) | 8 (8)
Skin laceration (Injury, poisoning and procedural complications) | 5 (10) | 10 (15)
Hypertension (Vascular disorders) | 7 (10) | 1 (2)
Blood pressure increased (Investigations) | 4 (9) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less